CLINICAL TRIAL: NCT00575172
Title: To Investigate Whether the Postprandial Blood Sugar Level as Achieved Using Ultrarapid-Acting Type Insulin Could Prevent Great Vessel Disorder in Japanese Type 2 Diabetic Patients.
Brief Title: Nippon Ultra-Rapid Insulin and Diabetic Complication Evaluation-Study (NICE-Study)
Status: Completed | Type: Observational
Sponsor: Osaka Saiseikai Nakatsu Hospital (Other)
Responsible Party: Osaka Saiseikai Nakatsu Hospital, NICE-study EBM center
Other Study IDs: UMIN0949; UMIN00000949
Record Dates: First submitted 2007-12-17; First posted 2007-12-18 (Estimated); Last update posted 2008-01-14 (Estimated); Status verified 2007-12

CONDITIONS: Diabetes Mellitus
Keywords: type2 diabetes mellitus; cardiovascular disease; macrovascular event
MeSH Terms: conditions — Diabetes Mellitus; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- U: Intensified insulin therapy with ultrarapid insulin-analogue (Insulin-Aspart)
- R: Intensified insulin therapy with human regular insulin

SUMMARY:
For the purpose of comparing efficacy of intensive therapy between 1) ultrarapid-acting type insulin (insulin aspart) and 2) conventional rapid-acting type insulin (R), a Multicenter Open Label Randomized Controlled Trial was planned in Japan using the occurrence of cardiovascular events in patients with diabetes, a high risk factor, as an index.

DETAILED DESCRIPTION:
A survey shows that the most frequently observed direct cause of death in diabetic patients is cardiovascular disorder. However, investigations and surveys such as DCCT, UKPDS and KUMAMOTO-study, etc. clarified that strict control of blood sugar level prevented development and progress of diabetic microangiopathy, but could not show a significant effect on great vessel disorder. Recently, the DECODA-study, DECODE-study and Honolulu-study have demonstrated that postprandial high blood sugar is involved in great vessel disorder. Therefore, possible prevention of great vessel disorder in diabetic patients is suggested by improving the postprandial blood sugar level as achieved using ultrarapid-acting type insulin, which has become available recently. Even with results in Europe and the US obtained, the life-style and incidence of complications in Japanese people are different, and there are many points that remain uncertain with respect to the direct application of foreign results to Japanese people. Therefore, in Japan also, it is necessary to conduct a large-scale clinical study and to establish high-level evidence using mainly Japanese people through hospitals having many patients.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are patients satisfying the following conditions 1) - 3).

  1. Outpatients and inpatients aged 20 years or more but younger than 85 years. Men or women.
  2. Patients with type 2 diabetes based on the diagnostic standard of the Japanese Diabetes Society
  3. No specific restriction on the current treatment. Patients having switched treatment are also accepted.

Exclusion Criteria:

1. Patients with type 1 diabetes
2. Patients with a past history of cerebral angiopathy (cerebral hemorrhage, cerebral infarction, transient cerebral ischemic attack, subarachnoid hemorrhage, etc.) within 6 months before giving consent
3. Patients with a past history of myocardial infarction within 6 months before giving consent
4. Patients planning to receive PTCA or CABG, or who had PTCA or CABG within 6 months before giving consent
5. Patients with coronary arteriopathy (angina pectoris, etc.) that requires treatment with β-blocker or calcium-antagonist
6. Patients with atrial fibrillation or atrial flutter
7. Patients with renal dysfunction (serum creatinine ≥ 3.0 mg/dL)
8. Patients with liver dysfunction (AST, ALT ≥ 100 IU/L)
9. Patients with a past history or suspected of having a malignant tumor within 5 years before giving consent
10. Pregnant or possibly pregnant patients
11. Other patients judged inappropriate for the study by the investigators (patients presenting difficulty in frequently receiving rapid-acting type insulin or ultrarapid-acting type insulin therapy, including patients' compliance with treatment)

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Japanese outpatients and inpatients aged 20 years or more but younger than 85 years. Men or women. Patients with type 2 diabetes based on the diagnostic standard of the Japanese Diabetes Society/American Diabetes Association. No specific restriction on the current treatment. Patients having switched treatment are also accepted.
Sampling Method: Probability Sample
Enrollment: 346 (Actual)
Dates: Start 2003-03; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Cardiovascular events 1)Sudden death 2)New development or recurrence of apoplexy or TIA 3)New development or recurrence of AMI or and angina pectoris 4)Newly developed ASO, amputation of leg due to ASO | five years

SECONDARY OUTCOMES:
1)Total mortality 2)Changes in the mean IMT of common carotid arteries 3)Changes in the pulse wave velocity (PWV) (rt & 1t baPWV), ABI | five years

CONTACTS AND LOCATIONS:
Overall Officials: Hideshi Kuzuya, M.D.,Ph.D, Study Chair — Higasiyama Takeda Hospital; Makoto Otoshi, MD.,Ph.D., Study Director — Ohtoshi Clinic; Haruo Nishimura, MD.,Ph.D., Principal Investigator — Osaka Saiseikai Nakatsu Hospital; Koji Maeda, MD., Principal Investigator — Maeda Clinic; Mitsuyo Shintani, MD.,Ph.D., Principal Investigator — Osaka Saiseikai Nakatsu Hospital
Locations (1):
- Osaka Saiseikai Nakatsu Hospital, Osaka, Osaka, Japan

REFERENCES:
- [Background] Nishimura H, Shintani M, Kouji M and Nice-study group J Saiseikai Nakatsu Hospital, 20, 216-220, 2003